CLINICAL TRIAL: NCT03395522
Title: One-arm, Multi-center, International Prospective Study to Assess the Efficacy of Medi-tate Temporary Implantable Nitinol Device (iTind) in Subjects With Symptomatic Benign Prostatic Hyperplasia (BPH)
Brief Title: Study to Assess the Efficacy of the iTind in Subjects With Symptomatic BPH
Acronym: MT-06
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medi-Tate Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-06
Record Dates: First submitted 2017-12-26; First posted 2018-01-10 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: BPH

STUDY DESIGN:
Intervention Model Description: device group only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device (Experimental): ITind device implant
  Interventions: Device: iTind

INTERVENTIONS:
Device: iTind — device implanted for 5-7 days

SUMMARY:
A total of up to 200 Symptomatic BPH subjects subjects will be enrolled into the study.

Study duration will be 12 months post implantation with a follow-up visits at Year 2 and Year 3.

DETAILED DESCRIPTION:
Primary Study Objective:

The study's primary objective is to assess the efficacy of the Medi-Tate iTind in subjects with symptomatic BPH by reduction of IPSS) (International Prostate Symptoms Score) score.

Secondary Study Objectives:

* To further evaluate the efficacy of Medi-Tate iTind as determined by increase of maximal urinary peak flow, satisfaction from the device and procedures, sex performance capabilities and ejaculation.
* Safety will be assessed by the rate of complications attributed to the Medi-Tate iTind and its implantation/retrieval procedures.

ELIGIBILITY:
Inclusion Criteria:

Subject signed informed consent prior to the performance of any study procedures.

* Male with symptomatic BPH: IPSS symptom severity score ≥ 10
* Peak urinary flow of < 12 ml/sec at flowmetry with minimum voided volume of at least 120 cc.
* Prostate volume 25 ml to 80 ml (as assessed by TRUS)
* Subject that is able to complete the study protocol
* Normal Urinalysis and urine culture.

Exclusion Criteria:

* Previous prostate surgery
* Prostate cancer
* Urethral stricture
* Bladder stones
* An active urinary tract infection.
* Obstructing median lobe demonstrated by IPP grade 3 (>1 cm) as assessed by TRUS.
* Neurological conditions potentially affecting voiding function.
* A post void residual (PVR) volume > 250 ml measured by ultrasound
* Previous diagnosis or treatment for Over Active Bladder
* Acute Urinary Retention
* Any anatomical or physiological condition that in the opinion of the investigator likely to impede successful completion of the study

Intra-Operation Exclusion:

• Obstructing median lobe or any other anatomical or physiological pathology that can interfere the device implantation as assessed by cystoscopy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male with symptomatic BPH
Enrollment: 149 (Actual)
Dates: Start 2018-02-18 (Actual); Primary Completion 2023-06-18 (Actual); Study Completion 2025-04-25 (Estimated)

PRIMARY OUTCOMES:
IPSS (International Prostate Symptoms Score) Responders Rate | at Month 6 Visit
  the Proportion (%) of Total IPSS Responders (3 points) Rate

SECONDARY OUTCOMES:
Total IPSS (International Prostate Symptoms Score) Score at | 6 months
  Change from Baseline to Month 6 in Total IPSS Score
Total IPSS(International Prostate Symptoms Score) Urinary Symptoms Score | 6 months
  Change from Baseline to Month 6 in Total IPSS Urinary Symptoms Score
Total SHIM (Sexual Health Inventory for Men ) Score | 6 months
  Change from Baseline to Month 6 in Total SHIM Score
Total ISI (Incontinence Severity Index ) Score | 6 months
  Change from Baseline to Month 6 in Total ISI Score
Total EJ-MSHQ ( Ejaculation- Male Sexual Health questionnaire) Score | 6 months
  Change from Baseline to Month 6 in Total EJ-MSHQ Score
Total Flow | 6 months
  Change from Baseline to Month 6 in Total Flow
Total residual urine | 6 months
  Change from Baseline to Month 6 in Total residual urine
Total Satisfaction Rate | 6 months
  Change from Baseline to Month 6 in Total Satisfaction Rate
IPSS QoL (Quality Of Life) score | 6 months
  Change from Baseline to Month 6 in IPSS QoL score
Recovery Success Rate | 1 month
  Quality of Recovery Success Rate

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Porpiglia, MD, Principal Investigator — San Orbessano
Locations (12):
- Sydney Adventist Hospital Clinical School of the University of Sydney, Sydney, Australia
- France (3):
  - Hospital Center University De Bordeaux, Bordeaux
  - Hôpital Cochin, Paris
  - Hôpital Privé des Côtes d'Armor, Plérin
- Germany (2):
  - University Hospital Frankfurt, Frankfurt
  - Medical center - University of Freiburg, Freiburg im Breisgau
- Italy (4):
  - AOU di Catanzaro, Catanzaro
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - San'Andrea Hospital, Rome
  - San Orbessano, Turin
- Clínica CEMTRO Ventisquero la Condesa, Madrid, Spain
- Cantonal Hospital St. Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No